CLINICAL TRIAL: NCT01799499
Title: A Prospective Open Label Comparative Dose Ranging Study Evaluating the Effect of Pre-TURBT Intravesical Instillation of Mitomycin C (MMC) Mixed With TC-3 Gel in Patients With Non Muscle Invasive Bladder Cancer (NMIBC)
Acronym: NMIBC TURBT HG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in the company clinical trials priority
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRE-TURBT-DR-PRO
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: Non Muscle Invasive Bladder Cancer; Intravesical instillation; Mitomycin C; Hydrogel; Reverse thermal gelation; Drug retention; Urinary Bladder Neoplasms; Carcinoma; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type Mitomycins; Mitomycin; Antibiotics, Antineoplastic; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions; Nucleic Acid Synthesis Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Alkylating Agents
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Carcinoma; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Neoplasms, Glandular and Epithelial

ARMS (3):
- Group A: 20 mg MMC mixed with 60cc TC-3 (Experimental): Group A: 20 mg MMC mixed with 60cc TC-3 hydrogel. (n=8)
  Interventions: Device: TC-3 hydrogel
- • Group B: 40 mg MMC mixed with 60cc TC-3 (Experimental): • Group B: 40 mg MMC mixed with 60cc TC-3 hydrogel (n=8)
  Interventions: Device: TC-3 hydrogel
- • Group C: 80 mg MMC mixed with 60cc TC-3 hydrogel (n=8) (Experimental): • Group C: 80 mg MMC mixed with 60cc TC-3 hydrogel (n=8)
  Interventions: Device: TC-3 hydrogel

INTERVENTIONS:
Device: TC-3 hydrogel
  Arms: Group A: 20 mg MMC mixed with 60cc TC-3
Device: TC-3 hydrogel
  Arms: • Group B: 40 mg MMC mixed with 60cc TC-3
Device: TC-3 hydrogel
  Arms: • Group C: 80 mg MMC mixed with 60cc TC-3 hydrogel (n=8)

SUMMARY:
This study is a prospective randomized open labeled dose ranging comparative study. Twenty four (24) patients with NMIBC who meet the inclusion/exclusion criteria will be recruited for the study following the initial diagnostic cystoscopy.

The investigators believe that this study is of importance on several aspects:

1. It evaluates a new mode of bladder instillation that may bypass the drawbacks of the current instillation mode.
2. If proved effective, this mode of treatment might save the need for TURBT performance and serve as a new mode of tumor ablation.
3. Even if proved partially effective, this mode of treatment will diminish tumors size and/or number, thus enable a more limited TURBT procedure.
4. This mode of treatment will enable immediate medical attendance to the patient's tumor recurrence without the waiting period (resulting from queues in the medical centers) for TURBT. This might improve the patient's prognostic outcome.
5. If this experimental treatment will prove to have a better ablative effect in comparison to the standard of care known in the art, this could be translated to a better prophylactic effect of tumor recurrence.
6. Finding the minimal, yet optimal, effective dose for tumor ablation and tumor recurrence prevention will enable us to reduce adverse effects of higher drug dosage.

DETAILED DESCRIPTION:
Non-muscle-Invasive Bladder cancer is mainly treated by tumor resection (Trans Urethral Resection - TUR), followed by series of intravesical instillations of prophylactic chemotherapeutic drugs such as Mitomycin C (MMC) or BCG. Unfortunately, this treatment approach is limited due to rapid dilution of the chemotherapeutic drug by the incoming urine and clearance by urination.

TheraCoat's core technology is based on a reverse thermal biodegradable gel (TC-3 Gel) (low viscosity at cold temperature (5°C) and gel appearance at body temperature)for drug retention in the urinary bladder.

Prior to instillation, the TC-3 Gel, in its liquid state, is mixed with MMC and instilled into the bladder by a standard catheter. Once inside the bladder, the gel solidifies and forms a drug reservoir. Upon contact with urine, the gel dissolves, release the drug slowly and is finally cleared out from the bladder.

Intravesical MMC instillation using TheraCoat's gel is expected to increase treatment efficiency due to prolongation of treatment duration and consequently improving bladder exposure to MMC.

Treatment Protocol - Immediately following baseline cystoscopy and tumor diagnosis and patient undergoes 6 weekly instillations followed by 2-4 weeks healing period.

1st Follow-Up Visit (Pre-Scheduled TURBT Visit): The patient will undergo a second cystoscopy to compare to baseline status. The patient will be followed-up for a period of 1 year as follows: 3,6,9,12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 21 years of age or older.
2. Patient has signed Informed Consent Form and is willing and able to abide by the protocol.
3. Single or multiple tumors (n≤7)
4. Naïve or Recurrent tumor
5. No prior history of HG and/or T1 and/or Tis
6. At least one Tumor ≥ 1mm as evaluated visually by the investigator
7. Largest tumor diameter ≤ 30mm as evaluated visually by the investigator
8. Cystoscopic appearance of papillary Low grade tumor
9. The patient had upper urinary tract evaluation in the previous year excluding urothelial carcinoma, hydronephrosis or Renal Cell Carcinoma or other renal cancers.
10. Good performance status (Karnofsky performance status 70% or greater).
11. No active urinary tract infection as confirmed by urine culture.
12. If the patient is a female of childbearing potential she is using an acceptable/effective method of contraception and has a negative pregnancy test at screening.

Exclusion Criteria:

1. Carcinoma In Situ (CIS).
2. Over 7 lesions
3. Lesion is larger than 30mm in diameter.
4. "High Grade" urine cytology.
5. Cystoscopic Appearance suspicious for HG and/or solid and/or Tis
6. histologic results of cold cup biopsy are indicative of HG tumor.
7. Tumor located in prostatic urethra.
8. Previous systemic chemotherapy or pelvic radiotherapy.
9. Pregnant or breastfeeding patient.
10. Previous treatment with BCG within the last 24 months.
11. The patient did not have at least 3 months cystoscopically confirmed tumor-free interval between the last tumor recurrence and screening.
12. Treatment with intravesical chemotherapy within the 3 last months.
13. The patient has/had any bladder tumor with histology other than TCC
14. Contraindication to MMC.
15. The patient has a history of urinary retention or a PVR≥250cc by bladder scan or ultrasound (PVR test may be repeated up to 3 times).
16. The patient has a bleeding disorder or a screening platelet count <50X109/L.
17. The patient has screening hemoglobin <10mg/dL.
18. The patient has a history of Acquired Immunodeficiency Syndrome or HIV positive.
19. The patient has a condition or a concurrent severe and/or uncontrolled medical or psychiatric disease (e.g. uncontrolled diabetes, compensated congestive heart failure (NYHA III and over), myocardial infarction within 6 months of study, unstable or uncontrolled hypertension or an active uncontrolled infection), which according to the PIs decision could compromise participation, compliance with scheduled visits and/or completion.
20. The patient participated in an investigational protocol within the past 90 days.
21. The patient has life expectancy of <3 years.
22. The patient had another malignancy or received therapy for any malignancy in the last five years except for:

    * Non-melanoma skin tumors
    * stage 0 (in situ) cervical carcinoma
    * prostatic carcinoma
23. The patient has documented vesica-ureteral reflux or an indwelling ureteral stent
24. The patient has the tumor in the bladder diverticulum

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ablative effect of pre-TURBT intravesical instillations with 20,40,80 mg of MMC mixed with 60cc TC-3 Hydrogel on bladder lesion(s) of NMIBC patients | 2 Years
  Cystoscopic and pathological effect (evaluated during TUR-BT visit) of pre-TURBT intravesical instillations with 20,40,80 mg of MMC mixed with 60cc TC-3 Hydrogel on bladder lesion(s) of NMIBC patients.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability rate. | 2 years
  Demonstration of Pre-TURBT TC-3 gel-MMC instillation safety and adverse event rate.Adverse events will be defined as any adverse change in health or side effect that occurs in the clinical trial participant while the patient is receiving the treatment or until the completion of the post-treatment follow-up cystoscopy.

OTHER OUTCOMES:
Comparison of the cystoscopic and pathological effect between the 3 groups. | 2 Years
  Comparison of the cystoscopic and pathological effect of pre-TURBT instillations between the 3 different dosages of MMC mixed with TC-3 Hydro-gel groups on bladder lesion(s).
one year tumor recurrence rate | 2 Years
  Comparison of one year tumor recurrence rate between the 3 treatment groups
PK level of MMC-C in blood | 1 Year
  Demonstration that blood levels of MMC following Pre-TURBT TC-3 gel-MMC instillation are below the toxic level (400ng/ml) known in the art for IV MMC administration

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital Nahariya, Nahariya, Israel